CLINICAL TRIAL: NCT01926327
Title: The Effects of Intraarticular Injection of Platelet-rich Plasma in Patients With Osteoarthritis of the Knee (in a Clinical Trial Phase III)
Brief Title: The Effect of Platelet-rich Plasma in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: royan-Bone-011
Record Dates: First submitted 2013-08-17; First posted 2013-08-20 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: PRP PRGF Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet reach plasma (Active Comparator): The patients with osteoarthritis who underwent PRP injection.
  Interventions: Biological: PRP injection
- placebo (Placebo Comparator): The patients with osteoarthritis who underwent Normal Saline injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PRP injection — Injection of PRP in patients with knee osteoarthritis.
  Arms: platelet reach plasma
Biological: Placebo
  Arms: placebo

SUMMARY:
Osteoarthritis is the most common type of arthritis. The prevalence of osteoarthritis of the knee has significantly elevated in the elderly population and youth due to age and sport activities respectively. Our aims to treat the knee osteoarthritis are including; reduce knee pain and improve its function; return patients to normal daily activities and reduce health care costs.

The current treatments which are already being used for osteoarthritis of the knee patients include:

1. Symptomatic therapy: conservative therapies, physiotherapy, analgesics and non-steroidal anti-inflammatory drugs.
2. Intra-articular injections of corticosteroids and hyaluronic acid.
3. Current Surgical Therapy: knee arthroplasty, osteotomy, arthrodesis and debridement.

As the low mitotic activity and lack of blood supply cause little ability for the articular cartilage to repair itself, so injection of platelet-rich plasma (PRP) has recently received much more attention due to its capacity to do self-healing in treatment of osteoarthritis of the knee.

PRP consists of several concentrated growth factors in platelets of autologous blood that are applied to the different parts of medicine such as reconstruction of damaged tissue. Although platelets are well-known to involve in the blood clots formation, but current studies have shown that they secrete many bio-proteins which attract macrophages, mesenchymal stem cells and osteoblasts to remove necrotic tissue in addition to participate in healing procedure.

This study is a prospective, randomized, controlled trial to assess The positive effects of platelet-rich plasma injection in 244 patients with osteoarthritis of the knee

DETAILED DESCRIPTION:
In this study all eligible patients (Based on the inclusion and exclusion criteria) were randomly allocated into two study groups by a Stratified Permuted Block randomization method: group A received platelet rich plasma, group B (control group) received only placebo.

All of the patients underwent a standard long protocol for knee osteoarthritis. All patients with grade II,III and IV of radiographic knee OA are selected. On average, in each instance, the amount of platelets in the peripheral blood is 4 to 6 times the baseline level.

Group A: 1-3 cc injection of placebo Group B: 1-3 cc injection of PRP All patients received monthly injection for 3 times.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years
2. Body mass index (BMI) ≤33 kg/m2
3. Grade 2And above imaging of osteoarthritis
4. History of knee pain or swelling should have at least 4 months

Exclusion Criteria:

1. treated with steroids and Anti-coagulant or anti-platelet aggregation
2. history of infectious, systemic diseases, Immune deficiency and coagulation disorders
3. Patients with Hb ≤11, Plt ≤ 150000
4. Varus > 10 , valgus > 10

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
pain | 3 months
  pain reduction by VAS scoring before injection of PRP and 3,6 and 12 months after last injection
physical activity | 3months
  physical activity of patients which is measured by WOMAC scoring , before injection of PRP& 3,6 and 12 months after last injection.
cartilage repair | 12months
  The repair of knee cartilage that is evaluated by MRI,before and 12months after injection.

SECONDARY OUTCOMES:
quality of life | 3months
  Evaluation the quality of life that is measured by SF36,before,3,6 and 12months after injection.
joint replacement | 12months
  Evaluation the need for joint replacement 12months after injection.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Nasser Aghdami, MD,PhD, Study Director — Head of Department of Regenerative Medicine Of Royan Institute & cell therapy center; Mohsen Emadedin, MD, Study Director — Orthoped scientist in Royan Institute; Ali Mirazimi Bafghi, MD, Principal Investigator — Regenerative Medicine Department of Royan Institute
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- See also: Related Info — http://royaninstitute.org